CLINICAL TRIAL: NCT05905198
Title: Programming Strategy of Variable Frequency Stimulation for Gait Impairments in Parkinson's Disease
Brief Title: Programming Strategy of VFS for Gait Impairments in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: K3438
Record Dates: First submitted 2023-02-22; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Parkinson's Disease; Deep Brain Stimulation; Gait Disorders, Neurologic
Keywords: Parkinson's disease; Deep brain stimulation; Variable frequency stimulation; Movement disorder; Freezing of gait; Crossover study
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic; Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFS-VFS (Experimental): This arm will experience HFS first during the crossover, and then VFS.
  Interventions: Device: Programming
- VFS-HFS (Experimental): This arm will experience VFS first during the crossover, and then HFS.
  Interventions: Device: Programming

INTERVENTIONS:
Device: Programming — programming the implanted DBS device to adjust the parameter and switch stimulation mode between Variable-Frequency settings and High-Frequency settings.

SUMMARY:
Variable Frequency Stimulation(VFS) is a stimulation pattern applied in Deep Brain Stimulation(DBS) therapy for Parkinson's disease(PD). Peking Union Medical College Hospital was the first centre conducting research on VFS. The studies in the past have resembled conclusion that VFS provides improvement not only in the major symptoms such as tremor and rigidity, but also in gait and balance disorder. However, the best programming strategy of VFS has not met agreement. The random-controlled double blinded crossover study is designed for participants who underwent DBS surgery in bilateral subthalamic nucleus for parkinson's disease. The investigators study several strategies on programming and observe the improvement of symptom to look for the best one. A 4-month follow-up is designed to observe a relatively long-term effectiveness of VFS. The study intends to gather more clinical evidence to guide further studies on VFS application.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (according to the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's Disease);
* 18-75 years of age;
* Hoehn & Yahr ≤ 3 (in best OFF-medication condition)；
* Implanted bilateral subthalamic nucleus DBS for over 1 year；
* gait Impairments in OFF-medication condition；
* High Frequency Stimulation provides significant improvement；
* in OFF-medication On-stimulation condition, capable of walking ≥ 10m.

Exclusion Criteria:

* mental disorder or dementia;
* Pregnant women, lactating mothers or women who are unable to take effective measures to prevent pregnancy;
* With other diseases that can affect walking distance, such as joint diseases of the lower body, spinal diseases, neuropathy, or serious heart or lung diseases;
* In severe health condition, such as diseases associated with heart or liver;
* Epilepsy;
* Lead off target;
* Unable to willingly sign Written informed Consent;
* Disagree or unable to cooperate with follow-up sessions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline 5m-Timed Up and Go test Time Result at 2 months. | Baseline, 2 months
  Conduct a TUG test with 5m range setting and measure the time cost
Change from Baseline 5m-Timed Up and Go test Time Result at 4 months. | Baseline, 4 months
  Conduct a TUG test with 5m range setting and measure the time cost

SECONDARY OUTCOMES:
Change from Baseline 5m-Timed Up and Go test Step Frequency at 2 months. | Baseline, 2 months
  Conduct a TUG test with 5m range setting and measure the step movement and calculate the step frequency
Change from Baseline 5m-Timed Up and Go test Step Frequency at 4 months. | Baseline, 4 months
  Conduct a TUG test with 5m range setting and measure the step movement and calculate the step frequency
Change from Baseline 5m-Timed Up and Go test Length at 2 months. | Baseline, 2 months
  Conduct a TUG test with 5m range setting and measure the length of each step
Change from Baseline 5m-Timed Up and Go test Step Length at 4 months. | Baseline, 4 months
  Conduct a TUG test with 5m range setting and measure the length of each step
Change from Baseline 5m-Timed Up and Go test Step Variation Coefficient at 2 months. | Baseline, 2 months
  Conduct a TUG test with 5m range setting and use the length of each step to calculate the difference coefficient
Change from Baseline 5m-Timed Up and Go test Step Variation Coefficient at 4 months. | Baseline, 4 months
  Conduct a TUG test with 5m range setting and use the length of each step to calculate the difference coefficient
Change from Baseline Movement Disorder Society Unified Parkinson's Disease Rating Scale part III score at 2 months. | Baseline, 2 months
  Conduct a Movement Disorder Society Unified Parkinson's Disease Rating Scale survey and record the score. Higher MDS UPDRS III score represents worse movement disorder symptoms.
Change from Baseline Movement Disorder Society Unified Parkinson's Disease Rating Scale part III score at 4 months. | Baseline, 4 months
  Conduct a Movement Disorder Society Unified Parkinson's Disease Rating Scale survey and record the score. Higher MDS UPDRS III score represents worse movement disorder symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Guo, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No